CLINICAL TRIAL: NCT02705248
Title: The Role of Insulin Resistance in Recurrent Miscarriage
Brief Title: Insulin Resistance in Recurrent Miscarriage
Acronym: IRRM
Status: Completed | Type: Observational
Sponsor: Ain Shams Maternity Hospital (Other)
Responsible Party: Principal Investigator, Nermine Essam El-Din Abdel-Salam, Dr Nermine Essam El-Din Abdel-Salam El-Serwi, Ain Shams Maternity Hospital
Other Study IDs: AinShamsMH 1
Record Dates: First submitted 2016-03-07; First posted 2016-03-10 (Estimated); Last update posted 2016-03-10 (Estimated); Status verified 2016-03

CONDITIONS: Insulin Resistance
MeSH Terms: conditions — Insulin Resistance

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- Group A: (Group A) case group: 40 pregnant females at 6- 13wks presenting with a history of recurrent pregnancy loss (two or more failed clinical pregnancies as documented by ultrasonography or histopathology examination according to the American Society of Reproductive Medicine) (ASRM, 2008).
- Group B: control group: 40 pregnant females at 6- 13wks with no history of abortion.

SUMMARY:
The objective of this study is to study the association between insulin resistance and recurrent spontaneous miscarriage (RSM).

DETAILED DESCRIPTION:
This a case-control study which was performed during the period from (December 2013) till (June 2014). Researcher had 80 participants presented to the outpatient clinic in Ain Shams University Maternity hospital; they were classified into two groups: (Group A) case group: 40 pregnant females at 6- 13wks presenting with a history of recurrent pregnancy loss (two or more failed clinical pregnancies as documented by ultrasonography or histopathology examination according to the American Society of Reproductive Medicine). (Group B) control group: 40 pregnant females at 6- 13wks with no history of abortion. They were selected according to inclusion and exclusion criteria:

* Inclusion criteria:

  1. Women in the child bearing period between 23-40 years.
  2. All patients were pregnant.
  3. The gestational age of both groups 6-13 weeks(1st trimester)
* Exclusion criteria:

  1. Patients with history of gestational diabetes.
  2. The patients on medication that could affect glucose metabolism at the time of the study (as metformin, Pioglitazone,rosiglitazone).
  3. Patients with other causes of recurrent abortion as (thyroid dysfunction, uterine anomalies, chromosomal abnormalities, antiphospholipid antibody syndrome).
  4. Patients with PCOS in the control group (they have insulin resistance).
  5. Obese patients (BMI >30).

The study was conducted after approval of the hospital ethical committee and a written consent was taken from all cases and controls participating in the study after full explanation. For all participants detailed history taking, full examination including body mass index was taken. The subjects were asked to go on a normal diet for 3 days prior to oral glucose tolerance test (OGTT). A fast for 8-10 h was required prior to sampling. A venous blood sample was drawn on the following morning from each subject to determine the concentrations of fasting glucose (FG) and fasting insulin (FI), afterwards subjects were required to drink a mixture of 75 g of pure glucose in 250 ml of water, venous blood samples were drawn again after 1, 2, and 3 h to determine the concentrations of glucose and insulin blood samples for determination of fasting glucose and fasting insulin after 8-10hours fasting and oral glucose tolerance test. Glucose concentration was determined using the hexokinase endpoint method; while insulin concentration was determined using the immunoluminescence method. The Immulite2000 Immunoassay Analyzer was used along with the necessary reagents. The homeostasis model assessment of insulin resistance index (HOMA-IR) for each subject was calculated as follows: [FI (U/ ml) ×FG (mmol/l)]/22.5.The larger the HOMA-IR, the more severe the degree of IR. HOMA-B, which represents the endocrine function of insulin, is calculated as 20× FI/ (FG-3.5). I 60 /I 0 represent the rate of 1-hour insulin to 1-hour glucose, and I60 / G60 represent the rate of 1-hour insulin increase to 1-hour glucose increase. Both values reflect the endocrine functions of B cells of the pancreatic gland. The area under the curve of glucose (AUCG) is equal to half of the FG plus

1-hour glucose, 2-hour glucose, and half of the 3-hour glucose. The area under the curve of insulin (AUCI) is also computed in this manner for insulin. The ratio AUCI/AUCG represents the rate of AUCI to AUCG, and the higher the rate, the more severe the degree of IR.

ELIGIBILITY:
Inclusion Criteria:

1. Women in the child bearing period between 23-40 years.
2. All patients were pregnant.
3. The gestational age of both groups 6-13 weeks(1st trimester)

Exclusion Criteria:

1. Patients with history of gestational diabetes.
2. The patients on medication that could affect glucose metabolism at the time of the study (as metformin, Pioglitazone,rosiglitazone).
3. Patients with other causes of recurrent abortion as (thyroid dysfunction, uterine anomalies, chromosomal abnormalities, antiphospholipid antibody syndrome).
4. Patients with PCOS in the control group (they have insulin resistance).
5. Obese patients (BMI >30).

Ages: 23 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: pregnant females in their first trimester (6- 13 weeks Gestational Age)
Sampling Method: Probability Sample
Enrollment: 80 (Actual)
Dates: Start 2013-12; Primary Completion 2014-06 (Actual); Study Completion 2016-03 (Actual)

PRIMARY OUTCOMES:
insulin resistance in patients with recurrent miscarriage | first trimester of pregnancy
  Insulin resistance was determined by measuring fasting Insulin, Fasting glucose, OGTT for all patients. the homeostasis model assessment of insulin resistance index (HOMA-IR) for each subject was calculated

CONTACTS AND LOCATIONS:
Overall Officials: Tarek M Tamara, Dr, Study Director — Ain Shams Maternity Hospital

IPD SHARING:
Plan to Share IPD: Undecided